CLINICAL TRIAL: NCT06973395
Title: The Effect of Individualized Nursing Interventions for Blood Glucose Variability Risk on Nursing Outcomes and Self-Management of Diabetes in Patients With Type 2 Diabetes
Brief Title: The Effect of Individualized Nursing Interventions on Glycemic Variability and Self-Management in Type 2 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Emel Bayraktar, Nursing Fundamentals Graduate Student, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AU-EBAYRAKTAR_001; Research Assistant PhD Student (Other: Ataturk University)
Record Dates: First submitted 2025-04-18; First posted 2025-05-15 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Type 2 diabetes; blood glucose variability; nursing diagnoses (NANDA); nursing interventions (NIC); nursing outcomes (NOC); diabetes self-management
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Methods; Educational Status

STUDY DESIGN:
Intervention Model Description: This research was planned as a randomized controlled screening study with repeated measurements and follow-ups, including pre-test, interim test and post-test, with experimental and control groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with nursing interventions applied (Experimental): Patient with type 2 diabetes.
  Interventions: Behavioral: Nursing interventions, education, and follow-up will be provided to Type 2 diabetes patients for blood glucose variability.
- Group without nursing interventions applied (No Intervention): Patient with type 2 diabetes. Only the survey will be applied to the control group.

INTERVENTIONS:
Behavioral: Nursing interventions, education, and follow-up will be provided to Type 2 diabetes patients for blood glucose variability. — Implementation of individual nursing interventions and provision of trainingIndividual nursing interventions will be applied to individuals with Type 2 diabetes regarding the risk of variability in blood glucose, and education and follow-up will be provided.
  Arms: Group with nursing interventions applied

SUMMARY:
Type 2 diabetes is a chronic disease with an increasing prevalence worldwide and in our country. In managing type 2 diabetes, the primary goal in the nursing process is to ensure blood glucose stability. In this regard, it is essential to provide individualized nursing interventions and diabetes management education to individuals. The Comprehensive Self-Management of Diabetes Scale can be used to determine individuals' level of diabetes management. Implementing systematic nursing interventions to maintain blood glucose stability and evaluating their impact on nursing outcomes and diabetes management are crucial. Although the NANDA, NIC, and NOC (NNN) system is used for this purpose, research in this area remains limited. There is a need for studies investigating the effects of individualized nursing interventions based on the NNN system on nursing outcomes and comprehensive self-management of diabetes in patients with type 2 diabetes who are at risk of blood glucose variability.

This study is planned as a randomized controlled trial with repeated measurements. The topic is original in terms of implementing individualized nursing interventions, providing education, and monitoring patients according to the NNN system to address the risk of blood glucose variability in patients with type 2 diabetes, as well as evaluating its impact on nursing outcomes and comprehensive self-management of diabetes. Another unique aspect of the study is that the effects of the interventions will also be assessed through laboratory results, including fasting blood glucose (FBG), postprandial blood glucose (PBG), HbA1c, height, weight, waist circumference, blood pressure, and pulse measurements.

This research aims to improve glycemic control, prevent potential complications of the disease, ensure patient safety, enhance the quality and satisfaction of nursing care, reduce additional treatment costs, and decrease diabetes-related morbidity and mortality.

If this study yields positive results, it will contribute to the widespread implementation of individualized nursing interventions using the NNN system to manage blood glucose variability risk, reduce diabetes-related health problems, ensure patient safety, and lower additional treatment costs. Furthermore, it is expected to guide clinical nurses, nurse researchers, and nurse managers in caring for individuals with type 2 diabetes, improve care quality and satisfaction, and support the planning of in-service training programs. From a healthcare institution perspective, it is anticipated to help reduce additional financial burdens and enhance care quality.

ELIGIBILITY:
Inclusion Criteria:

* Including the data of those aged 18-65,
* Those receiving oral antidiabetic treatment,
* Those who can use a smartphone and have internet access,
* Those who know how to write, read and speak Turkish,
* Those who do not have communication skills,
* Those who do not have a mental illness and are on psychiatric medication.

Exclusion Criteria:

* Individuals with liver and kidney failure, myocardial infarction, cerebrovascular accident and cancer
* Individuals receiving insulin treatment
* Individuals using steroid treatment will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Nursing outcomes level | Change in "Blood glucose level", "Hyperglycemia regimen", "Hypoglycemia regimen", "Diabetes management" and "Nutritional status" at 13 weeks
  Primary Outcome Measure 1:
  Name: Blood Glucose Level Time Frame: At weeks 1, 4, and 13 Description: Blood glucose level will be measured in mg/dL.
  Primary Outcome Measure 2:
  Name: Severity of Hyperglycemia Time Frame: At weeks 1, 4, and 13 Description: Severity of hyperglycemia will be evaluated based on blood glucose levels measured in mg/dL. Hyperglycemia level >135 mg/dL.
  Primary Outcome Measure 3:
  Name: Severity of Hypoglycemia Time Frame: At weeks 1, 4, and 13 Description: Severity of hypoglycemia will be evaluated based on blood glucose levels measured in mg/dL. (Hypoglycemia level <60 mg/dL) Primary Outcome Measure 4 Name: Nutritional Status Time Frame: At weeks 1, 4, and 13 Description: Nutritional status will be assessed using Body Mass Index (BMI), calculated as weight in kilograms divided by height in meters squared (kg/m²).
Comprehensive diabetes self-management performance level | "Change of comprehensive diabetes self-management at 13 weeks"
  The effect of individualized clinical interventions targeting the risk of blood glucose variability on the level of comprehensive diabetes self-management of Type 2 Diabetic Patients will be measured. Evaluation of changes in diabetes self-management behaviors using the Comprehensive Diabetes Self-Management Scale (CDSMS). Higher scores indicate better self-management.

CONTACTS AND LOCATIONS:
Overall Officials: Reva Balcı Akpınar, Prof. Dr., Study Director — Dean's Office of the Faculty of Nursing, Atatürk University
Locations (2):
- Turkey (Türkiye) (2):
  - Ataturk University Institute of Health Sciences, Erzurum, Turkey
  - Ataturk University, Erzurum, Turkey

IPD SHARING:
Plan to Share IPD: No